CLINICAL TRIAL: NCT05276128
Title: Evaluation of Potentially Bioactive Foods With Respect to Cardiometabolic- and Cognitive Test Variables
Brief Title: Effects of Plant Based Lipids on Glucose Regulation and Cognitive Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/658
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Diabete Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Lipids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WWB Reference (Other): White wheat bread (WWB) without lipid supplements. The effects of this high glycaemic product on postprandial glucose and insulin responses are well studied.
  Interventions: Dietary Supplement: lipids
- WWB 5g active lipids (Experimental): WWB supplemented with 5 g active lipids, and 10 g control lipids
  Interventions: Dietary Supplement: lipids
- WWB 10g active lipids (Experimental): WWB supplemented with 10g active lipids, and 5 g control lipids
  Interventions: Dietary Supplement: lipids
- WWB 15g active lipids (Experimental): WWB supplemented with 15g active lipids, and 0 g control lipids
  Interventions: Dietary Supplement: lipids
- WWB 15 g control lipids (Active Comparator): WWB supplemented with 15g control lipids
  Interventions: Dietary Supplement: lipids

INTERVENTIONS:
Dietary Supplement: lipids — Investigations of dose-response effects of 3 different doses of an bioactive plant based lipid consumed at breakfast, after overnight fasting. Total amounts of lipids in each test portion are 15g, and the lower doses are supplemented with a control lipid to sum upp to 15 g total lipids. A control product with15g control lipids and without active lipids is also included. The lipids are supplemented to a white wheat bread, corresponding to 50 g available starch. A White wheat bread portion without lipid supplementation is included as a well studied reference product.

SUMMARY:
The overall goal is to increase the knowledge that can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the primary purpose of this project is to evaluate effects in healthy humans on acute postprandial glucose regulation of plant based lipids. Due to the tight connection between cardiometabolic health and cognitive functions, a secondary issue is to investigate effects of test foods on cognitive test variables and mood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy subjects
* Between 20 and 40 years old
* Body mass index between 19-28 kg / m2),
* Consuming a non-vegetarian diet generally in line with the Nordic nutrition recommendations.

Exclusion Criteria:

* Fasting blood glucose concentration >6.1 mmol/L
* Known metabolic or gastrointestinal disorder (eg diabetes, high cholesterol, high blood pressure, IBS), or other disease that may affect the study results.
* Regular medication, except for long-term and stable medication for the lack or reduced production of thyroid hormone (eg Levaxin).
* Antibiotics or probiotics for at least four weeks before the start of the study,
* The use of tobacco products

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | 3 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Postprandial blood glucose responses

SECONDARY OUTCOMES:
Insulin responses | 3 hours. Fasting (time =0 minutes), 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Postprandial insulin responses
Mood variables | 60 minutes after start of test product, after 120 minutes and after 180 minutes
  Registration of subjective mood ratings (valence and activity) on 0-100 mm Visual Analogue Scales (VAS) at fasting and thereafter every hour until 180 min. Extremes of the sensations of the variables is at the two ends of the scales, i.e. 0 mm relates to the extrem of low senations sensations and 100 mm correspond to the highest sensation of the variables.
Appetite sensations | 3 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes
  Subjective sensations of hunger, satiety, and desire to eat are registered on 0-100 mm VAS scales. Extremes of the sensations of the variables is at the two ends of the scales, i.e. 0 mm relates to the extrem of low senations sensations and 100 mm correspond to the highest sensation of the variables.

OTHER OUTCOMES:
Cognitive test variable | 60 minutes after start of breakfast, after 120 minutes, and after 180 minutes
  Pilot study. Computerised test measuring aspects of selective attention, working memory and psychomotor reaction time

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Anne Nilsson, Lund, Välj...
  - The Human Trial Facility, Food Technology engineering and Nutrition, Lund University, Lund, Välj...

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make Individual Participant Data (IPD) and related data dictionaries available. The data will be published in a scientific journal as supplementary material simultaneously as the study results. The test persons names are coded and no individual participant can be identified.